CLINICAL TRIAL: NCT00470756
Title: Difference of Neuromuscular Activity in Infants and Toddlers With Foot Dorsiflexion Compare to Infants and Toddlers With Foot Plantarflexion
Brief Title: Forefoot Adduction (FFA) in Infants and Toddlers. Differences of Neuromuscular Activity.
Status: Suspended | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Naum Simanovski, Hadassah Medical Organization
Other Study IDs: SIM03-HMO-CTILL
Record Dates: First submitted 2007-05-06; First posted 2007-05-08 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-04

CONDITIONS: Forefoot Adduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- evertors, invertors
  Interventions: Other: mechanical triggering of peroneal activity

INTERVENTIONS:
Other: mechanical triggering of peroneal activity — mechanical triggering of peroneal activity

SUMMARY:
Every week we encounter with 5-8 pairs of worried parents of infants with forefoot adduction. Most of them usually need only reassurance and education how to manipulate the deformed foot. During the examination we usually use provocative maneuver to trigger peroneal activity. This manual stimulation usually reveals active eversion and dorsiflexion of the foot in most of the children, but not in all of them. Small part of the children reacts in opposite direction - instead of the typical eversion they demonstrate inversion and some plantar flexion of the foot. We have the impression that this subgroup of children improves the deformity slower and sometime less complete than most of the children. We did not find in the literature any description of this phenomenon. We postulate, that atypically reacting patients probably have different response due to abnormalities of neuromuscular balance between invertors-flexors and evertors-extensors muscle groups. This small subgroup of children may need more close follow-up and probably casting to speed up and secure the improvement of their deformity.

Study goals:

1. Evaluate ability of children with FFA to respond on mechanical triggering of peroneal activity

   1. The majority of the patients with standard reaction - foot dorsiflexion and eversion (evertors)
   2. The minority of the patients with nonstandard reaction - foot plantarflexion and inversion (invertors)
2. Evaluate randomly selected children from each group for character of muscular response on electrical stimulation (EMG) of calf muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Boys and girls between two months and one year old.
2. Non associated pathology.
3. Signing Informed consent.

Exclusion Criteria:

1. Unwillingness to sign informed consent.
2. Associated pathology

Ages: 2 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and toddlers with Forefoot adduction
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Naum Simanovski, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization., Jerusalem, Israel